CLINICAL TRIAL: NCT01039610
Title: A Single Center Four Part Study in Healthy Adult Subjects to Evaluate: the Safety, Tolerability and Pharmacokinetics of a Single Oral Dose and Repeat Escalating Oral Doses of GSK945237; the Effect of Linezolid on Hematology Safety Parameters; and the Effects of GSK945237 and Moxifloxacin on QTc.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Internal decision to progress alternate molecule with more preferable profile
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 107895
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Bacterial
Keywords: single dose; pharmacokinetics; GSK945237; tolerability; safety; antibiotics; linezolid; QTc; bacterial type II topoisomerase Inhibitors (BTI); moxifloxacin; repeat dose
MeSH Terms: conditions — Bacterial Infections | interventions — GSK945237; Linezolid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part A (Experimental): GSK945237 2400mg single dose
  Interventions: Drug: GSK945237; Drug: Placebo
- Part B Cohort 1 (Experimental): GSK945237 400 mg QD, 7 Days 4 subjects GSK945237:2 subjects Placebo
  Interventions: Drug: GSK945237; Drug: Placebo
- Part B Cohort 2 (Experimental): GSK945237 400 mg QD, 14 Days 4 subjects GSK945237:2 subjects Placebo
  Interventions: Drug: GSK945237; Drug: Placebo
- Part B Cohort 3 (Experimental): GSK945237 400 mg BID, 14 Days 4 subjects GSK945237:2 subjects Placebo
  Interventions: Drug: GSK945237; Drug: Placebo
- Part B Cohort 4 (Experimental): GSK945237 800 mg BID, 14 Days 9 subjects GSK945237:3 subjects Placebo
  Interventions: Drug: GSK945237; Drug: Placebo
- Part B Cohort 5 (Experimental): GSK945237 1200 mg BID, 14 Days 9 subjects GSK945237:3 subjects Placebo
  Interventions: Drug: GSK945237; Drug: Placebo
- Part B Cohort 6 (Experimental): GS945237 1600 mg QD, 14 Days 9 subjects GSK945237:3 subjects Placebo
  Interventions: Drug: GSK945237; Drug: Placebo
- Part C (Active Comparator): Linezolid 600 mg BID, 14 Days 9 subjects Linezolid:3 subjects Placebo
  Interventions: Drug: Placebo; Drug: Linezolid
- Part D (Active Comparator): 2 period crossover Period 1: Placebo 1 day; GSK945237 dose to be determined, 5 Days Period 2: Placebo 5 days; moxifloxacin 400 mg single dose
  16 subjects
  Interventions: Drug: GSK945237; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: GSK945237 — Dose detailed in Arm description
  Arms: Part A; Part B Cohort 1; Part B Cohort 2; Part B Cohort 3; Part B Cohort 4; Part B Cohort 5; Part B Cohort 6; Part D
Drug: Placebo — matching placebo tablet
Drug: Linezolid — 600 mg BID, 14 Days
  Arms: Part C
Drug: Moxifloxacin — 40 mg single dose
  Arms: Part D

SUMMARY:
GSK945237 belongs to the Bacterial Type II Topoisomerase Inhibitor (BTI) class of antibiotics. GSK945237 has demonstrated in vitro and in vivo activity against Gram positive [including methicillin resistant Staphylococcus aureus (MRSA)] and Gram-negative pathogens associated with respiratory tract, skin and soft tissue infections including isolates resistant to existing classes of antimicrobials. This study will be conducted in four (4) parts, with a single oral dose being explored in Part A (2400 mg) and repeat oral doses (b.i.d. and q.d.) being explored in Part B. Parts C and D will be optional evaluations of repeat oral doses of linezolid and a comparative evaluation of the effect of GSK945237 and moxifloxacin, respectively. Parts A and B will be single-blind, randomized, placebo-controlled, dose-rising (Part B only) studies of healthy subjects to evaluate the safety, tolerability and pharmacokinetics of GSK945237. The proposed doses range from 400 mg to 2400 mg. Part C will be a single-blind, randomized, and placebo-controlled repeat dose evaluation of 600 mg (b.i.d.) of linezolid. Part D will be a single-blind, randomized, placebo-controlled, two period crossover study. The proposed doses for Part D will be 1200 mg GSK945237 and 400 mg moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring. A subject with a non-clinically significant abnormality or laboratory parameters outside the reference range may be included only if the investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures or data interpretation.
* Male or female between 18 and 60 years of age.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented bilateral tubal ligation, hysterectomy, or bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until at least 90 days post-last dose.
* Body weight greater than 50 kg and BMI within the range 19 - 32 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any preexisting retinal condition or finding on baseline examination that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial or may interfere with interpretation of ophthalmologic safety results during the conduct of the trial.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins above the recommended daily intake herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 14 days prior to the first dose of study medication. By exception, the volunteer may take acetaminophen (< or equal to 2 grams/day) or ibuprofen (1600 mg/day) up to 48 hours prior to the first dose of study medication. However, the investigator and study team can review medication use on a case by case basis to determine if its use would compromise subject safety or interfere with study procedures or data interpretation.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* The subject has donated blood within 2 months prior to dosing and/or donated plasma within 1 week prior to dosing.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women, or an unwillingness of male subjects to use a condom and spermicide, in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of study medication administration and until 90 days after study medication administration.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* For Part C and Part D only: Contraindications to the use of linezolid or moxifloxacin, respectively as per the package insert [Avelox Product Information, 2008; Zyvox Product Information, 2008].

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessments, consisting of AEs, ECGs, vital signs, clinical laboratory tests. | duration of dosing
Plasma AUC(0-t), AUC(0-inf), Cmax, tmax, and t1/2 of GSK945237 | duration of dosing
Amount excreted in urine (Ae) and renal clearance of GSK945237 | duration of dosing
Saliva PK parameters | duration of dosing
QT interval and heart rate | duration of dosing
Change from baseline in QTc for GSk945237, moxifloxacin, and placebo | duration of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline